CLINICAL TRIAL: NCT02211781
Title: A Pilot Study of Dietary and Lifestyle Patterns Among Native Americans and Hispanics/Latinos in New Mexico at the Time of the Trinity Nuclear Test
Brief Title: Study of Diets and Way of Life of Native Americans and Hispanics in New Mexico During the Time of the Trinity Nuclear Test
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999914162; 14-C-N162
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05-21

CONDITIONS: Lifestyle; Diet; Ionizing Radiation Exposure
Keywords: Tribal Communities; Radiation; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective

SUMMARY:
Background:

- The National Cancer Institute has been studying health risks to people in New Mexico at the time of the first nuclear bomb test. This was called the Trinity nuclear test. It took place in 1945. Researchers want to also learn about Native Americans and Hispanics at that time. They want to learn about their way of life and their diets. This will give a more complete picture of the health risks to people in New Mexico in 1945.

Objectives:

* To learn about the activities and eating habits of Hispanic and tribal communities during the 1940s.
* To see if a group of Hispanic and Native Americans who were living in New Mexico in 1945 can be gathered.

Eligibility:

- Native American or Hispanic adults who were alive in 1945. They must know firsthand about the lifestyle and diet in New Mexico at that time.

Design:

* Participants will have 1 visit. They will be interviewed at a place like a library or office. They will answer questions about their lifestyle and diet around 1945. This will take up 60 90 minutes.
* Participants may agree to have their interviews taped. Their names will not be kept with their answers from the interviews.

DETAILED DESCRIPTION:
The evaluation of health risks among the public as a consequence of exposure to radioactive fallout from nuclear testing has been an important area of research for many years by investigators in the Radiation Epidemiology Branch (REB). As a result of the reputation of this group in the field of dose and risk assessment related to radioactive fallout, and the expertise of the National Cancer Institute (NCI) in cancer research, in 2007, U.S. Senator Jeff Bingaman (D, NM) sent a request to the NCI to evaluate the health risks to New Mexico residents from the first nuclear bomb test (named Trinity) that was conducted in 1945 in south-central New Mexico. The NCI responded in early 2008 with a preliminary evaluation of the radiation doses received by the residents of New Mexico. However, the evaluation made no special provisions for lifestyles and diets of tribal community members or Hispanics\Latinos which were a significant part of the population. Little is known about Native American and Hispanic\Latino lifestyles and diets in the mid-twentieth century, yet such data are necessary to produce a credible assessment of health risks to the state s population. For this reason, REB investigators did not publish the initial dose assessment in the peer-reviewed literature. Additionally, since statewide health records cannot be reconstructed in a meaningful way to determine excess disease rates, estimation of health risks in this population can only be projected (i.e., estimated) based on the magnitude and distribution of radiation doses received and the relationships between radiation dose and cancer risks observed in other populations. Since the preparation of the 2008 report, the REB exposure assessment models used to assess doses from radioactive fallout from other nuclear test sites have been improved and published in the peer-reviewed literature. The required improvements in the 2008 Trinity assessment that would support publication of the projected health risks includes sex- and age-dependent diet and lifestyle models for Native Americans and Hispanics\Latinos in New Mexico in the mid-1940s. We are proposing a pilot study to collect, via individual interviews, information on lifestyle and diet from up to 9 key informants of Native Americans and Hispanics\Latinos living in New Mexico who were alive at the time of the bomb (currently greater than or equal to 69 years old). This data will inform the design of a larger study, which will collect lifestyle and diet information from a series of targeted focus groups. The information acquired from these 9 individual interviews will be used to 1) determine the feasibility of assembling focus groups of members of tribal and Hispanic\Latino communities in New Mexico who were alive in 1945 at the time of the bomb and 2) provide lifestyle and diet information to be used for refining focus group interviewing tools.

ELIGIBILITY:
* Data Analysis Only

Ages: 75 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-08-01; Primary Completion 2014-08-01 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Diet and Lifestyle | September 2014

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Simon, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] Hellman A, Weislow OS, Twardzik DR, Fowler AK. Type C retrovirus activation and possible functions in the normal and tumor-bearing host. Cancer Res. 1979 Jul;39(7 Pt 2):2902-7. PMID 221111
- [Background] Schwerin M, Schonfeld S, Drozdovitch V, Akimzhanov K, Aldyngurov D, Bouville A, Land C, Luckyanov N, Mabuchi K, Semenova Y, Simon S, Tokaeva A, Zhumadilov Z, Potischman N. The utility of focus group interviews to capture dietary consumption data in the distant past: dairy consumption in Kazakhstan villages 50 years ago. J Dev Orig Health Dis. 2010 Jun;1(3):192-202. doi: 10.1017/S2040174410000243. PMID 24286002